CLINICAL TRIAL: NCT06609174
Title: Artificial Intelligence Electrocardiogram Enabled Mobile Device in Screening Families for Dilated Cardiomyopathy (The AI-SCREENDCM Decentralized Clinical Trial Pilot Study)
Brief Title: AI-SCREENDCM Decentralized Clinical Trial - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Naveen L. Pereira, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 24-006256
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Cardiomyopathy
Keywords: Artificial Intelligence
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- First degree relatives (Experimental): Subjects who are first-degree relatives of patients with DCM
  Interventions: Diagnostic Test: KardiaRx ECG Screening and AI interpretation of ECG
- DCM (Dilated Cardiomyopathy) Patients (Experimental): Subjects who are diagnosed with DCM (dilated cardiomyopathy).
  Interventions: Diagnostic Test: KardiaRx ECG Screening and AI interpretation of ECG

INTERVENTIONS:
Diagnostic Test: KardiaRx ECG Screening and AI interpretation of ECG — The Kardia 6-lead device is an ambulatory, wireless device that connects to a smartphone. The KardiaRx App processes the signal acquired from the Kardia device into a real-time ECG. ECG will be interpreted by an AI algorithm

SUMMARY:
The purpose of this study is to assess the feasibility and impact of screening FDR of DCM probands using a mobile ECG with the ability to transmit the ECG for cloud-based AI analysis to detect reduced left ventricular ejection fraction (LVEF). This protocol will examine the impact of incorporating the screening AI enhanced ECG into standard of care recommendations.

ELIGIBILITY:
Inclusion Criteria (Proband)

* Male or female age ≥ 18 years
* Confirmed diagnosis of DCM determined at the discretion of the treating physician and defined as LVEF ≤ 45% at any time during the clinical course of the patient
* Must have at least one living ≥ 18 years FDR
* Able to provide informed consent

Inclusion Criteria (FDR)

* Male or female age ≥ 18 years who are first-degree relatives of patients with DCM
* Proband has provided informed consent
* FDR able to provide informed consent
* Access to a smartphone or digital tablet with cellular data or Wi-Fi access

Exclusion Criteria (Proband)

* DCM attributed to any other secondary form of cardiomyopathy per the investigator's determination
* Proband has previously informed FDR to undergo cardiac screening
* Ischemic cause of reduced LVEF

  * evidence of myocardial infarction, inducible ischemia or chest pain on stress testing in absence of coronary angiogram to rule out ischemic disease
  * history of acute coronary syndromes (STEMI, NSTEMI or unstable angina) revascularization or ≥75% stenosis of either left main or LAD or ≥75% stenosis of 2 major epicardial vessels on angiogram
* Moderate or greater primary valvular abnormality not due to underlying cardiomyopathy
* Congenital structural heart disease
* Severe and untreated or untreatable hypertension
* Cardiomyopathy due to acute or reversible conditions; examples include tachyarrhythmias, thyroid disorders, iron overload
* Any secondary cause of reduced LVEF such as pregnancy, myocarditis, amyloidosis, sarcoidosis, exposure to toxins including alcohol, substance abuse or chemotherapeutic drug
* (CPC Participants only) Home address outside of traveling range

Exclusion Criteria (FDR)

* Previously informed about cardiac screening or has completed cardiac screening by TTE
* Previously diagnosed with reduced LVEF
* (CPC Participants only) Home address outside of traveling range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Number of First-Degree Relatives to complete the AI-ECG | Baseline
  Measured by the number of complete transmissions from the Kardia 6-lead device to the AI-ECG algorithm.
Number of First-Degree relatives to complete cardiac screening | Baseline
  The following screening procedures will be considered a valid cardiac screening attempt:
  * Scheduled or Completed TTE
  * Scheduled or completed clinician visit for the purposes of generating a cardiac evaluation

SECONDARY OUTCOMES:
Number of subjects with an Left Ventricular Ejection Fraction ≤ 45% | Baseline
  Left Ventricular Ejection Fraction will be determined by AI-ECG

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Pereira, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No